CLINICAL TRIAL: NCT06453694
Title: A Pilot Randomized Trial of Efgartigimod Alfa for the Treatment of Incident Moderate to Severe Acute Optic Neuritis
Brief Title: Efgartigimod for the Treatment of Acute Optic Neuritis
Acronym: PET-AON
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anastasia Vishnevetsky, MD, MPH (Other)
Collaborators: argenx (Industry)
Responsible Party: Sponsor-Investigator, Anastasia Vishnevetsky, MD, MPH, Attending Physician in Neurology, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: pet-aon-001
Record Dates: First submitted 2024-05-30; First posted 2024-06-12 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Optic Neuritis
Keywords: Optic neuritis; Inflammatory optic neuropathy; Myelin Oligodendrocyte Glycoprotein Antibody Disease (MOGAD); Neuromyelitis Optica Spectrum Disorder (NMOSD); Multiple Sclerosis
MeSH Terms: conditions — Optic Neuritis; Neuromyelitis Optica; Multiple Sclerosis | interventions — efgartigimod alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efgartigmod alfa (Active Comparator): 10 patients will receive efgartigimod alfa
  All participants will receive standard of care high dose corticosteroids for 3 days with a prednisone taper over 3 weeks.
  Interventions: Drug: Efgartigimod Alfa
- Placebo (Placebo Comparator): 10 patients will receive placebo.
  All participants will receive standard of care high dose corticosteroids for 3 days with a prednisone taper over 3 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Efgartigimod Alfa — 2,016 mg will be administered subcutaneously by a healthcare provider on Day 0 and Day 3 of the trial.
  Rescue therapy with therapeutic plasma exchange will be given to any participant based on the results of Day 7 evaluation.
  Other Names: Vyvgart Hytrulo
  Arms: Efgartigmod alfa
Drug: Placebo — Subcutaneous injection of placebo will be administered by a healthcare provider on Day 0 and Day 3 of the trial.
  Rescue therapy with therapeutic plasma exchange will be given to any participant based on the results of Day 7 evaluation.
  Arms: Placebo

SUMMARY:
The goal of this pilot clinical trial is to test efgartigimod alfa against placebo in adults with first-time optic neuritis (optic nerve inflammation). The main questions it aims to answer are:

* Is it feasible to use efgartigimod alfa for optic neuritis?
* Is it feasible to run a larger trial testing efgartigimod alfa in optic neuritis?
* Does efgartigimod alfa work better than placebo in improving how quickly and how much vision returns?

Participants will:

* have their vision and blood tested
* be asked questions about their vision
* will receive standard of care treatment with steroids regardless of whether they are receiving efgartigimod alfa or not
* will have periodic visits over 6 months

DETAILED DESCRIPTION:
This study is designed as a pilot, single-site, randomized, placebo-controlled, 2-arm, parallel-group clinical trial comparing efgartigimod alfa in addition to standard of care (IV steroids with a standardized oral taper) to standard of care with placebo, with an option for rescue therapy with plasma exchange for all participants in the case of poor therapeutic response.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Adults aged 18 years or older
4. Diagnosed with a first episode of optic neuritis, based on clinical presentation (i.e. typical features such as pain with eye movements, color vision changes, subacute presentation, and visual acuity loss) and confirmed by contrast enhancement or T2 hyperintensity of the optic nerve on MRI brain or orbits using a 1.5T MRI scanner or greater
5. Onset of optic neuritis-related vision changes (does not include headache, eye pain, or pain with eye movements), as defined by decreased visual acuity, subjectively reported blurred vision, or optic nerve enhancement on MRI brain or orbits, within 10 days (inclusive) of enrollment. If optic neuritis is bilateral, then enrollment must occur within 10 days of vision changes in the first affected eye.
6. Best-corrected high contrast visual acuity (HCVA) in the worse affected eye on the Early Treatment Diabetic Retinopathy Study (ETDRS) eye chart of logMAR 0.48 (20/60) or worse.
7. For females of reproductive potential: negative urine or serum pregnancy test at screening or use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 8 weeks after the end of efgartigimod administration
8. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner

Exclusion Criteria:

1. Current pregnancy or lactation
2. Known allergic reactions or intolerance to efgartigimod, methylprednisolone, prednisone, or gadolinium or any of their components
3. Known diagnosis of optic neuropathy preceding the current episode of optic neuritis
4. Evidence of a systemic disease other than MS, NMOSD, or MOGAD that might be associated with the optic neuritis
5. Receiving systemic immunomodulatory or immunosuppressive therapy at the time of enrollment or planned receipt within 3 weeks of treatment. Initiation of immunotherapy more than 3 weeks after the second dose of efgartigimod is not an exclusion criterion and is permitted.
6. Known diagnosis of CNS demyelinating disease (MS, NMOSD, MOGAD) prior to present attack.
7. Any visually-significant ocular pathology (i.e. retinal problems, cataracts, glaucoma etc.) in the affected eye that led to known best-corrected visual acuity deficits in participants prior to onset of optic neuritis. Congenital color-blindness is not disqualifying.
8. Alternative explanation for visual changes detected on fundoscopic exam and slit lamp examination.
9. Enrollment in another clinical study involving an investigational treatment given within 2 months of enrollment in the present study.
10. Contraindication to MRI or plasma exchange
11. Has received >3 days of high-dose steroids (IV or PO) for the treatment of the current episode of acute optic neuritis by the time of randomization. Randomization may occur at the latest on the next day after completion of 3rd dose of steroids.
12. Known HIV disease or common variable immunodeficiency
13. History of malignancy unless considered cured by adequate treatment with no evidence of recurrence for ≥1 year before the first administration of IMP. Adequately treated participants with the following cancers may be included at any time:

    1. Basal cell or squamous cell skin cancer
    2. Carcinoma in situ of the cervix
    3. Carcinoma in situ of the breast
    4. Incidental histological finding of prostate cancer (TNM stage T1a or T1b)
14. Clinically significant uncontrolled active or chronic bacterial, viral, or fungal infection
15. Clinically significant recent major surgery (within 1 month of screening), or intends to have surgery during the study
16. Any conditions or circumstances that in the opinion of the investigator may put the participant at undue risk, confound the results of the study, or otherwise make the participant unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | 2 years
  Number of enrolled participants per month
Study Adherence Rate | 2 years
  Proportion of randomized participants who receive both doses of assigned study intervention, attend all assigned study visits, and complete at least the high contrast visual acuity, low contrast visual acuity, and Pelli-Robson assessments at all visits
Change in high contrast visual acuity for effect size and standard deviation estimation | 1 month
  Difference in change in high-contrast visual acuity from baseline to 1 month between groups
Change in low contrast visual acuity for effect size and standard deviation estimation | 1 month
  Difference in change in low contrast visual acuity (LCVA) (# of letters seen at 2.5% illumination) from baseline to 1 month between groups

SECONDARY OUTCOMES:
Retention rate | 2 years
  Percentage of enrolled subjects who remain in the study and do not voluntarily withdraw
Screen failure rate | 2 years
  Percentage of participants who fail screening
Pre-screen failure rate | 2 years
  Percentage of participants who fail pre-screening
Drug adherence rate | 2 years
  Percentage of randomized participants who receive 2 full doses of their assigned study intervention
Full improvement in visual acuity (high contrast) | 30 days
  Proportion of participants with full improvement in high contrast visual acuity
Full improvement in visual acuity (low contrast) | 30 days
  Proportion of participants with full improvement in low contrast visual acuity
Personal maximal improvement (high contrast) | 30 days
  Proportion of participants with personal maximal improvement in high contrast visual acuity (defined as individual final visual acuity at 6 months)
Personal maximal improvement (low contrast) | 30 days
  Proportion of participants with personal maximal improvement in high contrast visual acuity (defined as individual final visual acuity at 6 months)
Improvement in high contrast visual acuity at 3 months | 3 months
  Difference in change in high contrast visual acuity from baseline to 3 months between groups
Improvement in high contrast visual acuity at 6 months | 6 months
  Difference in change in high contrast visual acuity from baseline to 6 months between groups
Rescue treatment | Day 7
  Number and proportion of patients in each arm requiring rescue treatment
Difference in change in low contrast visual acuity from baseline to 6 months between groups | 3 months
  Difference in change in low contrast visual acuity (# of letters seen at 2.5% illumination) from baseline to 3 months between groups
Difference in change in low contrast visual acuity from baseline to 6 months between groups | 6 months
  Difference in change in low contrast visual acuity (# of letters seen at 2.5% illumination) from baseline to 6 months between groups
The number and proportion of participants with low contrast visual acuity of 0 | 30 days
  The number and proportion of participants with low contrast visual acuity of 0
Contrast sensitivity | 6 months
  Difference in change in Pelli-Robson contrast sensitivity score (# of letters seen at 2.5% illumination) from baseline to each assessment time point between groups
Color Vision | 6 months
  Difference in change in Hardy-Rand-Rittler color vision score from baseline to each assessment time point between groups. Scores range from 0 (lowest) to 6 (highest).
Visual fields | 6 months
  Difference in change in Humphrey Visual fields score from baseline to each assessment time point between groups. Data derived from automated perimetry are continuous and expressed in decibels. The mean deviation calculated from a Humphrey Visual Field analyzer (24-2 fast paradigm) represents the difference between an individual's test performance and the performance of a normally-sighted control of the same age.
Vision Related Quality of Life | 6 months
  National Eye Institute Visual Functioning Questionnaire (VFQ-25) scores at baseline, 1 month, 3 months, and 6 months in each arm. Scores range from 0 = worst to 100 = best
Efgartigimod safety measures | 6 months
  Frequency and type of overall adverse events, treatment-related adverse events, and serious adverse events

OTHER OUTCOMES:
Number and proportion of patients enrolled within 3, 5, 7, and 10 days of visual symptom onset | Day 0
  Number and proportion of patients enrolled within 3, 5, 7, and 10 days of visual symptom onset
Contrast enhancement | Day 0
  Number and proportion of patients enrolled with contrast enhancement of the optic nerves on MRI
Median duration (in days) from onset of blurry vision or visual acuity change to randomization | Day 0
  Median duration (in days) from onset of blurry vision or visual acuity change to randomization
Median duration (in days) from onset of eye pain or headache to randomization | Day 0
  Median duration (in days) from onset of eye pain or headache to randomization
Number and proportion of overall participants with each diagnosis | Day 30
  Number and proportion of overall participants with a final diagnosis of AQP4+ NMOSD, seronegative NMOSD, MOGAD, MS-related optic neuritis, idiopathic acute optic neuritis, or other diagnosis
Proportion amongst screened and recruited participants with HCVA of each visual acuity severity | Day 0
  Proportion amongst screened and recruited participants with HCVA worse than logMAR 0.48 (20/60), logMAR 0.7 (20/100), and logMAR 1 (20/200)
Retinal nerve fiber layer (RNFL) thickness at 1 month between groups | 1 month
  Retinal nerve fiber layer (RNFL) thickness at 1 month between groups
Retinal nerve fiber layer (RNFL) thickness at 3 months between groups | 3 months
  Retinal nerve fiber layer (RNFL) thickness at 3 months between groups
Retinal nerve fiber layer (RNFL) thickness at 6 months between groups | 6 months
  Retinal nerve fiber layer (RNFL) thickness at 6 months between groups
Ganglion cell layer (GCL) thickness at 1 month between groups | 1 month
  Ganglion cell layer (GCL) thickness at 1 month between groups
Ganglion cell layer (GCL) thickness at 3 months between groups | 3 months
  Ganglion cell layer (GCL) thickness at 3 months between groups
Ganglion cell layer (GCL) thickness at 6 months between groups | 6 months
  Ganglion cell layer (GCL) thickness at 6 months between groups

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Vishnevetsky, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No